CLINICAL TRIAL: NCT06620835
Title: Optimization of Treatment With Brigatinib in Patients With Advanced NSCLC Harboring an ALK Rearrangement by LAT at the Time of Best Response: A Multicenter Open Phase Two Trial (OPTALK)
Brief Title: Trial for Local Ablative Treatment (LAT) Optimization in Patients With Advanced Non-Small Cells Lung Cancer (NSCLC) Presenting an Anaplastic Lymphoma Kinase (ALK) Rearrangement Treated by Brigatinib
Acronym: OPTALK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Optalk GFPC 07-2023; 2024-A00356-41 (Other: ANSM/CPP)
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: NSCLC
Keywords: NSCLC; Lung cancer; ALK rearrangement; gene mutation
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Hematologic Tests; Pregnancy Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical Trial population (Experimental): All advanced non-small cell lung cancer (NSCLC) patients with ALK rearrangements treated with brigatinib in first line of non-curable setting will be screened.
  If the disease assessment done between 3 to 9 months after initiation of brigatinib shows:
  * a tumor response or stabilization (according to RECIST 1.1)
  * a disease which meets the definition of an oligometastatic disease (five metastatic lesions or less and a maximum of two lesions per organ)
  * all tumor targets are accessible to a local ablative therapy (confirmed by an expert panel of clinicians before inclusion): surgery, stereotactic radiosurgery (SRS), For liver, adrenal, or other metastases, percutaneous thermal ablation will be accepted.
  Eligible patients will benefit from local ablative therapy with continuation of brigatinib.
  Interventions: Biological: Blood samples for Hematology; Biological: Blood samples for Chemistry; Biological: Blood sample for liver function tests; Biological: Pregnancy test; Procedure: Tumour assessment; Procedure: Local Ablative Therapy (LAT)

INTERVENTIONS:
Biological: Blood samples for Hematology — Complete blood count will include erythrocytes, neutrophils, eosinophils, basophils, lymphocytes, monocytes, platelets, leukocytes, hemoglobin, hematocrit.
Biological: Blood samples for Chemistry — Clinical chemistry will include serum electrolytes (sodium, potassium, calcium, corrected calcium for hypoalbuminemia), creatinine, CrCl with local formula, and fasting blood glucose.
Biological: Blood sample for liver function tests — Laboratory tests to assess liver function will include Aminotransferase Alanine (ALAT), Aminotransferase Aspartate (ASAT), Phosphatase Alkaline (ALP), Gamma-glutamyl Transferase (GGT), total and conjugated bilirubin.
Biological: Pregnancy test — Pregnancy test will be performed in women of childbearing potential, including women who have had a tubal ligation. Childbearing potential is defined as not having undergone surgical sterilization, hysterectomy, and/or bilateral oophorectomy or not being postmenopausal (≥12 months of amenorrhea). Urine pregnancy tests will be based on the measurement of β-Human Chorionic Gonadotropin (HCG). If a urine pregnancy test is positive, it must be confirmed by a serum pregnancy test. Urine pregnancy tests will be performed at screening.
Procedure: Tumour assessment — Tumor assessment according to the RECIST v1.1 include the following radiological evaluation: thoracic CT scan, brain MRI or CT scan (MRI is preferred), abdominopelvic scan, PET-CT scan mandatory and at the Investigator's discretion, if needed bone scintigraphy and chest X-ray.
Procedure: Local Ablative Therapy (LAT) — Local Ablative Treatment (LAT) (stereotactic body radiotherapy, surgery, thermal ablation)

SUMMARY:
The goal of this clinical trial is to learn if the treatment by systemic Brigatinib (ALUNBRIG®) associated to local ablative therapy (LAT) treatment is improved if administered when the brigatinib works best in participants presenting an advanced non-small cells lung cancer with an ALK gene anomaly (this anomaly produces a defective protein that is responsible for the multiplication of cancer cells).

This clinical trial is expected to involve 45 participants in several sites in France.

Advanced non-small cell lung cancer (NSCLC) participants with ALK rearrangements treated with brigatinib in first line of non-curable setting will be screened.

If the disease assessment done between 3 to 9 months after initiation of brigatinib shows:

* a tumor response or stabilization (according to RECIST 1.1)
* a disease which meets the definition of an oligometastatic disease (five metastatic lesions or less and a maximum of two lesions per organ)
* all tumor targets are accessible to a local ablative therapy (confirmed by an expert panel of clinicians before inclusion): surgery, stereotactic radiosurgery (SRS). For liver, adrenal, or other metastases, percutaneous thermal ablation will be accepted.

Participants will be asked to visit the clinic:

* for eligibility criteria assessment prior to LAT
* for LAT
* every 8 weeks for checkups and tests the first year after LAT
* and then every 12 weeks, for a maximum period of 3 years.

Eligible patients will benefit from local ablative therapy with continuation of brigatinib.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at diagnosis.
* Stage 3 non eligible for chemoradiotherapy or stage 4 NSCLC, histologically or cytologically confirmed NSCLC.
* Tyrosine Kinase Inhibitor (TKI) treatment naïve.
* ALK rearrangements identified by a validated technique (either Immunohistochimy (IHC), fluorescence in situ hybridization (FISH) or Ribonucleic Acid (RNA)seq, in tissue or liquid biopsy)
* Stable disease or response after initiation brigatinib treatment (at least 3 to 9 months) according to RECIST 1.1
* At least one site of residual site for LAT (ie. participant should not have a complete response)
* Oligometastatic disease (five metastatic lesions or less and a maximum of two lesions per organ) de novo or induced
* Eligible for local ablative treatment possible (either alone or combined): surgery, minimally invasive form of surgical radiosurgery (Stereotactic Radio Surgery (SRS)) (18 to 20 Gy in single fraction) or radiotherapy (SBRT) (27 to 54 Gy in 3 fractions or 45 to 50 Gy in 5 fractions), radiofrequency or cryotherapy (=thermoablation)
* An Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2.
* Life expectancy above 12 weeks as assessed by treating investigator.
* Brain metastases at inclusion are allowed if asymptomatic
* No history of other malignant tumor during the previous 5 years, except for adequately treated carcinomas (in situ cervical carcinoma, basal cell carcinoma, squamous cell skin carcinoma) and low-grade localized prostate cancer (Gleason <6).
* Adequate organ function, as demonstrated by laboratory results prior to the first administration of study treatment: normal hepatic function (bilirubin ≤1.5 x upper limit of normal (ULN), alanine aminotransferase (ALA T) and aspartate aminotransferase (ASAT) ≤2.5 x ULN or ≤5 x ULN in case of liver metastases), renal function (calculated creatinine clearance (CrCl, using local formula) above 45 ml/mn), normal hematological function (absolute neutrophil count

  ≥1.5 x 109/L and/or platelets ≥100 x 109/L, hemoglobin ≥8 g/dL), normal coagulation function (International Normalized Ratio (INR) or prothrombin time ≤1.5 x ULN and activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) ≤1.5 x ULN unless the patient is receiving anticoagulant therapy)
* For patients of childbearing potential: Women of childbearing potential should use effective non-hormonal contraception during treatment with brigatinib and for at least 4 months following the final dose. Men with female partners of childbearing potential should use effective contraception during treatment and for at least 3 months after the last dose of brigatinib.
* Signed informed consent to participate in the study
* Affiliation with or benefit from French social security

Exclusion Criteria:

* NSCLC without known ALK rearrangements
* Neuroendocrine tumor (even in case of mixed tumors).
* Uncontrolled and untreated superior cava syndrome.
* Unstable symptomatic brain metastases despite corticosteroid
* Leptomeningeal, pericardial, pleural and mesenteric lesions, lymphangitic spread (any tumoral lesions not amenable to definitive local therapy). Peri tumoral lymphangitic spread around a tumor, but limited to a lobe, may be treated by surgery).
* Serious concurrent conditions during the previous 6 months (severe or unstable angina pectoris, coronary or peripheral artery bypass graft of <6 months, class 3 or 4 congestive heart failure, ischemic stroke, grade ≥2 peripheral neuropathy, psychiatric or neurological disorders that may interfere with the patient's understanding of the study or with his/her informed consent.
* Severe or non-controlled systemic diseases deemed incompatible with the protocol.
* Severe infections within 4 weeks prior to inclusion, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Psychological, family, social, or geographical factors that may interfere with the monitoring of the patient as defined by the protocol.
* Any protected person (legal person protected by legal protection [guardianship, tutorship], person deprived of liberty, pregnant woman, breastfeeding woman, and minor).
* Patients who participated in other concomitant studies unless observational and received study therapy or used an investigational device within 4 weeks prior to start of study treatment
* Known allergies or adverse reactions to the study drugs
* Lung function not compatible with surgery or radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) centrally assessed | From the start date of treatment up to the disease progression as per central reading or for a maximum of 3 years.
  PFS is defined as the time from Brigatinib initiation until tumor progression or death from any cause according to RECIST v1.1, evaluated by the expert panel.
  Radiological evaluation of the target lesions(s) will be performed at the following time points: Screening, then every 8 weeks during the first year then every 12 weeks thereafter.
  An expert panel of blinded clinicians will anonymously review the radiological evaluations and confirm/infirm the Investigator's assessment. Each Investigator must provide all the documents necessary to assess the various endpoints.
  Progression occurring before 2 years will be considered for the endpoint. Patients alive without progression will be censored at the last radiological assessment.

SECONDARY OUTCOMES:
Progression free survival (PFS) locally assessed | From the start date of treatment up to the disease progression as per local reading or for a maximum of 3 years.
  PFS is defined as the time from Brigatinib initiation until tumor progression or death from any cause according to RECIST v1.1, evaluated by the investigators.
  Radiological evaluation of the target lesions(s) will be performed at the following time points: Screening, then every 8 weeks during the first year then every 12 weeks thereafter.
  If a Computed Tomography (CT) scan for tumor assessment is performed in a Positron Emission Tomography (PET) scanner or CT scanner, the CT acquisition must be consistent with the standards for a full-contrast diagnostic CT scan.
  Response will be assessed by the Investigator at each center using RECIST v1.1. Assessments should be performed by the same evaluator, if possible, to ensure internal consistency across visits.
  Progression occurring before 2 years will be considered for the endpoint. Patients alive without progression will be censored at the last radiological assessment.
Overall survival (OS) | From the start of treatment until death or lost of follow-up or for a maximum of 3 years
  Overall survival defined as the time from Brigatinib initiation until death or lost of follow up.
  Patients alive will be censored at the date of last news or data cutoff. The patient's status (dead, alive or censored) will be determined at the same time points as PFS (Screening, then every 8 weeks during the first year then every 12 weeks thereafter) in order to evaluate OS. In addition, OS will be determined during the Post-study Follow-up Period via in-person or phone contact every 3 months.
Median PFS | From the start of treatment until death or lost of follow-up or for a maximum of 3 years
  Median PFS defined as the time from Brigatinib initiation until death or lost of follow up.
  Patients alive without progressive disease will be censored at the date of last news or data cutoff.
Safety and tolerability | From the enrolment of the participant up to until 90 days after the last administration of radiotherapy or until 60 days after the last surgery / thermal ablation
  Safety and tolerability : proportion of patients with any adverse event (AE), serious AEs (SAEs) and all AEs of grade ≥3 according to the National Cancer Institute (NCI) Common terminology criteria for adverse events (CTCAE) v5.0 criteria.
  Participants will be monitored for AEs from the time the informed consent form is signed until 90 days after the last administration of radiotherapy or until 60 days after the last surgery / thermal ablation. Safety assessments may include monitoring of any or all of the following parameters: clinical symptoms, laboratory, pathological, radiological or surgical findings, results of physical examination, or results of other tests and/or procedures.
  Any later SAE, i.e. occurring after the end of the reporting period, which is considered to be related to the trial intervention(s) or to the research (protocol required diagnostic procedures and examinations carried out during the research) must be reported without any limitation in terms of deadline.
Duration of Treatment (DOR) | From the start date of treatment up to stop date of treatment or for a maximum of 3 years
  Duration of treatment, defined as the time from the first Brigatinib treatment administration until the date of last treatment administration. Dates of first and last treatment administration will be recorded for each treatment to calculate the duration of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard AULIAC, Principal Investigator — Centre Hospitalier Intercommunal de Créteil Service Pneumologie; Isabelle MARTEL LAFAY, Principal Investigator — Centre Léon Bérard Service Radiothérapie
Locations (27):
- France (27):
  - CHU de Brest, Brest
  - Centre François Baclesse, Caen
  - CH Métropole-Savoie, Chambéry
  - Hôpital Louis Pasteur, Colmar
  - Pneumologie Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Georges-François Leclerc, Dijon
  - CH Annecy, Épagny
  - Polyclinique de Blois, La Chaussée-Saint-Victor
  - CHD les Oudaries, La Roche-sur-Yon
  - CHU Dupuytren, Limoges
  - Centre Leon Bérard, Lyon
  - Hôpital Nord, Marseille
  - CHRU de Nancy, Nancy
  - CLCC Antoine Lacassagne, Nice
  - CHU de Nîmes, Nîmes
  - CHU Orléans, Orléans
  - Hôpital Tenon, Paris
  - CHU de Bordeaux Haut Lévêque, Pessac
  - CHU Rennes, Hôpital Pontchaillou, Rennes
  - CHU Ponchailloux, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Pneumologie CHU St Etienne, Saint-Etienne
  - CHU de la Réunion, Saint-Pierre
  - Centre Paul Strauss, Strasbourg
  - HIA St Anne, Toulon
  - CH Bretagne Atlantique, Vannes
  - Centre Hospitalier de Villefranche sur Saone, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Undecided